CLINICAL TRIAL: NCT00132197
Title: Treatment of Patients With Chronic Functional Disorders. A Randomized Controlled Trial of Specialized Treatment Compared to Usual Care.
Brief Title: Treatment of Patients With Longstanding Unexplained Health Complaints
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus County, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20052
Record Dates: First submitted 2005-07-19; First posted 2005-08-19 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Somatization Disorder
Keywords: Functional somatic symptoms; Cognitive behavioral therapy; somatization disorder; SF-36; cost-effectiveness; Medically unexplained symptoms
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 1. Specialised treatment includes cognitive groups therapy in 9 modules of 3,5 hours within 3½ months, in all 31,5 hours, consultancy over the phone to the patients' GPs and tuition in groups headed by an experienced social worker. Detailed treatment manuals are worked out separately for each module. Experienced psychotherapists (clinical psychologists and psychiatrists), who also function as consultants, will do the treatment. The Ph.D.-student functions as co-therapist.
Procedure: Recommendation of care (letter to general practitioner [GP]) — After the diagnostic assessment the patient does not receive any treatment offers at the research clinic, but the patient and the GP will be informed about the diagnosis, and the GP will receive advice on further treatment possibilities.

SUMMARY:
The purpose of this study is to determine the effect of specialized treatment (including cognitive therapy, social counselling and a recommendation letter to the patients' primary care physician) on the functional level, emotional problems, and use of health care in patients with chronic medically unexplained symptoms.

DETAILED DESCRIPTION:
Medically unexplained or functional somatic symptoms are complaints, which are not attributable to any verifiable, conventionally defined disease, or which cannot adequately be supported by clinical or para-clinical findings.

Functional somatic symptoms are common in the population and in all clinical settings, both in primary and secondary care. The disorders range from mild, transitory cases, which are difficult to delimit in relation to normality, to severe chronic cases with multiple symptoms from different organ systems.

Chronic multiple functional somatic symptoms often cause frustration for both GPs and patients due to lack of availability of specialized treatment offers. Patients may have a high use of health care, and their social and functional level is low. In Denmark, patients with chronic multiple functional somatic symptoms account for at least 10% of the early retirement pensions each year.

Diverse interventions have been effective in the management and treatment of patients with functional disorders. Care recommendation letters for the GPs have both helped reduce the patients' use of health care and improved their level of physical functioning. Randomized controlled trials (RCT) have shown that cognitive behavioral treatment (CBT) has effect on specific patient groups with functional disorders. Through a combination of cognitive behavioral therapy, social counselling and recommendation letters, it is possible to offer patients with chronic functional somatic symptoms a presumably effective and cost-effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple somatic symptoms from several organ systems, without adequate medical explanation.
* Moderate to severe influence on daily life.
* The disorder's functional component can easily be separated from a possible well-defined chronic somatic illness.
* No lifetime-diagnosis of psychoses, bipolar affective disorder or depression with psychotic symptoms (International Classification of Diseases [ICD-10]: F20-29, F30-31, F32.3, F33.3)
* The condition must have been present for at least 2 years.
* Patients of Scandinavian origin who understand, read, write and speak Danish.

Exclusion Criteria:

* No informed consent.
* An acute psychiatric disorder that demands other treatment, or if the patient is suicidal.
* Abuse of narcotics or alcohol and (non-prescribed) medicine.
* Pregnancy.
* Current industrial injury case or other action for damages.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2005-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Physical health measured with The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) (aggregate score of the scales physical functioning, bodily pain and vitality) | Measured at baseline and months 4 (end of treatment), 10 and 16

SECONDARY OUTCOMES:
Psychosocial effect measures: Social level of functioning, emotional disorders, coping strategies measured with relevant sub-scales from the SF-36, WHO-DAS II, CSQ, Symptom Checklist SCL, Whiteley-7 | Measured at baseline and months 4 (end of treatment), 10 and 16
Use of health care measured by information from the National Patient Register, the Psychiatric Central Register, the National Health Service Register and The Danish Medicines Agency | Measured for a period of one year prior to referral (baseline) and a period of one year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Per Fink, Dr.Med.Sc., Study Director — The Research Clinic for Functional Disorders, Aarhus University Hospital
Locations (1):
- Per Fink, Aarhus C, Denmark

REFERENCES:
- [Derived] Schroder A, Rehfeld E, Ornbol E, Sharpe M, Licht RW, Fink P. Cognitive-behavioural group treatment for a range of functional somatic syndromes: randomised trial. Br J Psychiatry. 2012 Jun;200(6):499-507. doi: 10.1192/bjp.bp.111.098681. Epub 2012 Apr 26. PMID 22539780
- See also: Related Info — http://www.functionaldisorders.dk